CLINICAL TRIAL: NCT07134907
Title: The Efficacy and Safety of Qianweitai (Silodosin Capsule) Compared to Tamsulosin in the Treatment of Benign Prostaic Hyperplasia (BPH) -A Multicenter, Prospecive, Randomized, Investigator-Blind, Positive-Controlled Study
Brief Title: The Efficacy and Safety of Qianweitai (Silodosin Capsule) Versus Tamsulosin in the Treatment of BPH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Huilun Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NM-22-A-001-YJ-001
Record Dates: First submitted 2025-08-14; First posted 2025-08-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: BPH (Benign Prostatic Hyperplasia)
Keywords: Benign Prostatic Hyperplasia; Qianweitai; Tamsulosin; Lower Urinary Tract Symptoms
MeSH Terms: conditions — Prostatic Hyperplasia; Lower Urinary Tract Symptoms | interventions — silodosin

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Qianweitai (Experimental): Patients orally take Qianweitai (silodosin capsule), 4mg/capsule, 1 capsule/time, bid, after breakfast and dinner).
  Interventions: Drug: Silodosin
- Tamsulosin (Active Comparator): Patients orally take tamsulosin hydrochloride capsules (1 tablet each time, once daily).
  Interventions: Drug: Tamsolusin

INTERVENTIONS:
Drug: Silodosin — Silodosin is an α1A-adrenergic receptor antagonist which can relax the smooth muscle of bladder and prostate, relieve the dynamic obstruction of bladder outlet, and improve the lower urinary tract symptoms caused by BPH. The instruction of Silodosin Capsule (Qianweitai®) is 4mg/capsule，1 capsule/time, bid, after breakfast and dinner.
  Other Names: Qianweitai
  Arms: Qianweitai
Drug: Tamsolusin — Tamsulosin is an α1A-adrenergic receptor blocker which has used in treatment of BPH for few years. The instruction of Tamsulosin Capsule is 1 tablet at a time, 1 time a day.
  Other Names: Harnal
  Arms: Tamsulosin

SUMMARY:
The goal of this clinical trial is to learn if Qianweitai (QWT, silodosin capsule) works to treat BPH/LUTS in male adults. It will also learn the safety about QWT. The main questions it aims to answer are:

1. Whether QWT is non inferior to tamsulosin in the reduction of IPSS total score？
2. Dose QWT have other advantages in the improvement of LUTS?

Participants will:

1. Orally take QWT twice daily or tamsulosin once daily for 12 weeks.
2. Visit the clinic at week 1、 2、4、8 and 12 for checkups and tests.

DETAILED DESCRIPTION:
This trial is designed as two stages: screening period, treatment and follow-up period.

Screening period (days -28 to 0): After signing the informed consent form, the subjects entered into the screening period, and made a 24-hour urination diary and screening examination.

Treatment and Follow-up period: eligible patients were randomly assigned to 2 groups according to 1: 1 and received Tamsulosin or Silodosin or for 12 weeks. During the treatment period, the subjects' diaries were recorded according to the requirements of the scheme, and they were followed up at 1 week (7±2 days), 2 weeks (14±3), 4 weeks (28±5 days), 8 weeks (56±7 days) and 12 weeks (84±10 days). During the visit, relevant scale scores and laboratory examinations were performed, and the occurrence of adverse events during the follow-up was recorded to evaluate the safety.

ELIGIBILITY:
Inclusion Criteria:

1. Male Subjects aged 60 ～ 80 years, clinically diagnosed as benign prostatic hyperplasia.
2. Has an IPSS score ≥ 8 points at Screening and Baseline.
3. Has a 4 ≤ Qmax ≤ 15 ml/s when urination volume > 150 ml.
4. Has a prostate volume (PV) ≥ 30 ml by ultrasound examination.
5. Subjects who can read, understand, and complete the research questionnaire.
6. Subjects willing to participate voluntarily in this clinical trial, give informed consent and sign informed consent.

Exclusion Criteria:

1. Subjects with prostate cancer or other malignant tumors.
2. Subjects have serum tPSA > 10ng/ml, or 4 ≤ tPSA ≤ 10ng/ml while fPSA/tPSA < 0.16 times.
3. Subjects suffered from other diseases causing dysuria, such as bladder neck spasm, urethral stricture, neurogenic bladder dysfunction, etc.
4. Subjects have suffered from acute urinary retention, or complicated with gross hematuria, urinary tract infection, bladder stones, secondary upper urinary tract hydronephrosis, urinary incontinence, renal insufficiency and other Subjects that researchers believe meet the surgical indications.
5. Subjects have undergone prostate surgery, microwave therapy, urethral dilatation or acute urinary retention catheterization or other invasive procedures.
6. Subjects have residual urine volume (PVR) > 100ml, or those who may have urinary retention and need catheterization.
7. Subjects who took α receptor blockers, traditional Chinese medicine or botanical drugs for treating BPH within two weeks before participating this clinical trial.
8. Subjects who take 5α reductase inhibitor or other antiandrogen therapy drugs within half a year before participating this clinical trial.
9. Subjects who need to take drugs prohibited in this study or adopt prohibited treatment methods during treatment.
10. Subjects who Complicated with severe cardiovascular and cerebrovascular diseases, respiratory diseases, blood diseases, liver and kidney diseases.
11. There are significant abnormalities in clinical or laboratory examination indexes of patients, such as ALT and AST ≥ 2.5 times of the upper limit of reference value, creatinine (Scr) > 1.5 times of the upper limit of reference value, or poor blood glucose control (fasting blood glucose FPG ≥ 10 mmol/L).
12. Subjects who are allergic to the drugs or ingredients used in the test definitely.
13. Any otherSubjects in the opinion of researchers is not suitable for inclusion.

Ages: 60 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2022-07-18 (Actual); Primary Completion 2024-07-09 (Actual); Study Completion 2024-07-09 (Actual)

PRIMARY OUTCOMES:
International Prostate Symptom Score（IPSS） | week 12
  Changes of IPSS scores at the 12th week of treatment compared with baseline scores.

SECONDARY OUTCOMES:
International Prostate Symptom Score（IPSS） total score | 1, 2, 4 and 8 weeks
  Changes of IPSS scores at 1, 2, 4 and 8 weeks after treatment compared with baseline
IPSS storage subscore | 1, 2, 4 and 8 weeks
  Changes of IPSS storage subscore at 1, 2, 4 and 8 weeks after treatment compared with baseline
IPSS voiding subscore | 1, 2, 4 and 8 weeks
  Changes of IPSS voiding subscore at 1, 2, 4 and 8 weeks after treatment compared with baseline
IPSS total score severity | week 12
  Proportion of patients with IPSS total score severity decreased by at least one grade at 12 weeks. The scores of the scale were divided into three grades: mild (0-7), moderate (8-19) and severe (20-35).
Quality of life (QoL) score | 4, 8 and 12 weeks
  Changes in scores at 4, 8 and 12 weeks of treatment compared with baseline.The scores of the scale ranged from 0 to 6. The higher the score, the more severe the symptoms are.
Maximum urinary flow rate (Qmax) | week 12
  The change of Qmax at the 12th week of treatment compared with baseline.
Residual urine volume (PVR) | week 12
  The change of PVR at the 12th week of treatment compared with baseline.
Prostate specific antigen (PSA) | week 12
  The change of PSA at the 12th week of treatment compared with baseline.
Prostate volume (PV) | week 12
  Changes of PV at 12 the 12th week of treatment compared with baseline.
Responder rate | week 12
  Responder rate is defined as the proportion of patients whose IPSS total score decreased by ≥ 25% and Qmax increased by ≥ 30% compared with baseline value after treatment.
Proportion of patients with BPH clinical progression | week 12
  Clinical progress is defined as the first occurrence of one of the following two conditions during the trial:
  1. Acute urinary retention (AUR);
  2. Clinical diagnosis requires surgical treatment of BPH.

CONTACTS AND LOCATIONS:
Overall Officials: Shan Chen, Principal Investigator — Beijing Tongren Hospital
Locations (6):
- China (6):
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Wuhan Center Hospital, Wuhan, Hubei
  - Wuhan No.1 Hospital, Wuhan, Hubei
  - The Second Affiliated Hospital of Suzhou University, Suzhou, Jiangsu
  - Beijing Tongren Hospital, Capital Medical University, Beijing
  - Ciivil Aviation General Hospital, Beijing